CLINICAL TRIAL: NCT03882060
Title: The Effect of Recombinant Human Erythropoietin on the Postoperative Neurologic Outcome in Pediatric Moyamoya Disease Patients - A Double Blind Randomized Controlled Trial
Brief Title: Effect of Recombinant Human EPO on the Postoperative Neurologic Outcome in Pediatric Moyamoya Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1812-165-999
Record Dates: First submitted 2019-03-12; First posted 2019-03-20 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Moyamoya Disease; Pediatrics; Cerebrovascular Disorders
MeSH Terms: conditions — Moyamoya Disease; Cerebrovascular Disorders | interventions — Erythropoietin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rHuEPO (Experimental): recombinant human erythropoietin 500 U/kg IVS x 3 times Preoperative day (12-24 hour before surgery) During surgery Postoperative day (12-24 hour after surgery)
  Interventions: Drug: erythropoietin
- Control (Placebo Comparator): Normal saline 50mL x 3 times Preoperative day (12-24 hour before surgery) During surgery Postoperative day (12-24 hour after surgery)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: erythropoietin — Recombinant human erythropoietin (500 U/kg IVS x 3 times) is administrated to increase the neovascularization after revascularization surgery.
  Other Names: rHuEPO
  Arms: rHuEPO
Drug: Normal saline — Control group, no intervention.
  Other Names: Control
  Arms: Control

SUMMARY:
This study evaluates the effect of recombinant human erythropoietin (rHuEPO) on the neovascularization of pediatric moyamoya disease patients. rHuEPO will be administrated during perioperative period of the first revascularization surgery. Primary outcome (Incidence of Good postoperative MCA territory revascularization by cerebral angiography) will be evaluated after 3-6 month of revascularization surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Moyamoya patients scheduled for the first revascularization surgery

Exclusion Criteria:

* Hypersensitivity or contraindication to rHuEPO
* History of Unstable hypertension, Hypertensive encephalopathy, Thrombosis
* Primary intracerebral hemorrhage (ICH), Subarachnoid hemorrhage (SAH), Arterio-venous malformation (AVM), Cerebral aneurysm, or cerebral neoplasm
* History of seizure
* Hemoglobin >16 mg/dl
* Prolonged PT (PT > 15.5 seconds, PT INR > 1.2) or Prolonged aPTT (> 40 seconds)
* Thrombocytopenia (platelet count < 100,000/microL), Thrombocytosis (platelet count > 400,000/microL), Neutropenia (absolute neutrophil count (ANC) < 1500/microL)
* Abnormal kidney function (Creatinine> 2.0 mg/dl, History of dialysis)
* Abnormal hepatic function (aspartate transaminase> 80 unit/L, alanine aminotransferase> 80 unit/L)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative <12 month Angiogenesis | <12 month after revascularization operation
  Incidence of Good postoperative MCA territory revascularization by cerebral angiography or MRI (3 grade: good, fair, poor)

SECONDARY OUTCOMES:
Short-term postoperative outcome: Incidence and number of the postoperative transient ischemic attack (TIA) within 1 week | up to 1 week
  Incidence and number of the postoperative transient ischemic attack (TIA) within 1 week (yes or no)
Short-term postoperative outcome: Adverse neurologic event | within the 1st postoperative hospital stay, up to 1 year
  seizure, increased intracranial pressure, cerebral infarct, hematoma, reoperation (yes or no)
Short-term postoperative outcome: Other postoperative complications | within the 1st postoperative hospital stay, up to 1 year
  e.g. Circulatory failure/arrest, Respiratory failure/arrest, Infection (yes or no)
Short-term postoperative outcome: ICU stay (days) | within the 1st postoperative hospital stay, up to 1 year
  ICU stay (discharge criteria: Stable V/S + Consciousness)
Short-term postoperative outcome: Total hospital stay (days) | within the 1st postoperative hospital stay, up to 1 year
  Total hospital stay (discharge criteria: Stable V/S + no progressive Sx)
Effect of rHuEPO on perioperative erythropoiesis: Total intraoperative and perioperative transfusion requirements (mL/kg) | within the 1st postoperative hospital stay, up to 1 year
  Total intraoperative and perioperative transfusion requirements (mL/kg)
Effect of rHuEPO on perioperative erythropoiesis: Perioperative Hemoglobin, Hematocrit, serum EPO level | within the 1st postoperative hospital stay, up to 1 year
  Perioperative Hemoglobin, Hematocrit, serum EPO level
Effect of rHuEPO on perioperative erythropoiesis: GFR, BUN, Creatinine | within the 1st postoperative hospital stay, up to 1 year
  GFR, BUN, Creatinine level
Postoperative <12 month neurologic outcome: Clinical outcomes (4 grade): Excellent, Good, Fair, Poor | Outpatient clinical visit, Usually Postoperative 3~6 month, up to 1 year
  Clinical outcomes (4 grade): Excellent, Good, Fair, Poor
Postoperative <12 month neurologic outcome: Brain Perfusion MRI (2 grade): Favorable, Unfavorable | Outpatient clinical visit, Usually Postoperative 3~6 month, up to 1 year
  Brain Perfusion MRI (2 grade): Favorable, Unfavorable
Long-term neurologic outcome: Clinical outcomes (4 grade): Excellent, Good, Fair, Poor | Outpatient clinical visit, Usually Postoperative 12~18 month, up to 2 years
  Clinical outcomes (4 grade): Excellent, Good, Fair, Poor
Long-term neurologic outcome: Brain MRI/A or Brain perfusion MRI | Outpatient clinical visit, Usually Postoperative 12~18 month, up to 2 years
  Brain MRI/A or Brain perfusion MRI (2 grade): Favorable, Unfavorable
Long-term neurologic outcome: Cognitive function assessed by Korean Wechsler Intelligence Scale for Children-Ⅳ (K-WISC-Ⅳ) | Outpatient clinical visit, Usually Postoperative 12~18 month, up to 2 years
  Cognitive function assessed by Korean Wechsler Intelligence Scale for Children-Ⅳ (K-WISC-Ⅳ, has 4 domaines: Verbal Comprehension Index, Perceptual Reasoning Index, Working Memory Index, Processing Speed Index > final score is calculated from T-score)
Preoperative Cerebral angiography: Suzuki grade, Bilateral involvement | Before up to 1 year
  Cerebral angiography: Suzuki grade(1-6), Bilateral involvement (yes/no)
Preoperative Brain MRI/A or Brain Perfusion MRI | If the preoperative w/u is not completed before recruitment, up to 1 week
  Brain MRI/A or Brain Perfusion MRI (2 grade): Favorable, Unfavorable
Preoperative Hemoglobin, Hematocrit, serum EPO level | If the preoperative w/u is not completed before recruitment, up to 1 week
  Preoperative Hemoglobin, Hematocrit, serum EPO level
Preoperative information: Homozygous RNF213 | If the preoperative w/u is not completed before recruitment, up to 1 week
  Homozygous RNF213

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hong JM, Lee SJ, Lee JS, Choi MH, Lee SE, Choi JW, Lim YC. Feasibility of Multiple Burr Hole With Erythropoietin in Acute Moyamoya Patients. Stroke. 2018 May;49(5):1290-1295. doi: 10.1161/STROKEAHA.117.020566. Epub 2018 Apr 6. PMID 29626135
- [Background] Malla RR, Asimi R, Teli MA, Shaheen F, Bhat MA. Erythropoietin monotherapy in perinatal asphyxia with moderate to severe encephalopathy: a randomized placebo-controlled trial. J Perinatol. 2017 May;37(5):596-601. doi: 10.1038/jp.2017.17. Epub 2017 Mar 9. PMID 28277490
- [Background] Kimakova P, Solar P, Solarova Z, Komel R, Debeljak N. Erythropoietin and Its Angiogenic Activity. Int J Mol Sci. 2017 Jul 13;18(7):1519. doi: 10.3390/ijms18071519. PMID 28703764
- [Background] Aljaaly HA, Aldekhayel SA, Diaz-Abele J, Karunanayka M, Gilardino MS. Effect of Erythropoietin on Transfusion Requirements for Craniosynostosis Surgery in Children. J Craniofac Surg. 2017 Jul;28(5):1315-1319. doi: 10.1097/SCS.0000000000003717. PMID 28582302
- [Background] Wu YW, Mathur AM, Chang T, McKinstry RC, Mulkey SB, Mayock DE, Van Meurs KP, Rogers EE, Gonzalez FF, Comstock BA, Juul SE, Msall ME, Bonifacio SL, Glass HC, Massaro AN, Dong L, Tan KW, Heagerty PJ, Ballard RA. High-Dose Erythropoietin and Hypothermia for Hypoxic-Ischemic Encephalopathy: A Phase II Trial. Pediatrics. 2016 Jun;137(6):e20160191. doi: 10.1542/peds.2016-0191. Epub 2016 May 2. PMID 27244862
- [Background] Bang OY, Fujimura M, Kim SK. The Pathophysiology of Moyamoya Disease: An Update. J Stroke. 2016 Jan;18(1):12-20. doi: 10.5853/jos.2015.01760. Epub 2016 Jan 29. PMID 26846756
- [Background] Kim T, Oh CW, Bang JS, Kim JE, Cho WS. Moyamoya Disease: Treatment and Outcomes. J Stroke. 2016 Jan;18(1):21-30. doi: 10.5853/jos.2015.01739. Epub 2016 Jan 29. PMID 26846757
- [Background] Yoo YC, Shim JK, Kim JC, Jo YY, Lee JH, Kwak YL. Effect of single recombinant human erythropoietin injection on transfusion requirements in preoperatively anemic patients undergoing valvular heart surgery. Anesthesiology. 2011 Nov;115(5):929-37. doi: 10.1097/ALN.0b013e318232004b. PMID 22027622
- [Background] Kim SK, Cho BK, Phi JH, Lee JY, Chae JH, Kim KJ, Hwang YS, Kim IO, Lee DS, Lee J, Wang KC. Pediatric moyamoya disease: An analysis of 410 consecutive cases. Ann Neurol. 2010 Jul;68(1):92-101. doi: 10.1002/ana.21981. PMID 20582955
- [Background] Kim JH, Jung JH, Phi JH, Kang HS, Kim JE, Chae JH, Kim SJ, Kim YH, Kim YY, Cho BK, Wang KC, Kim SK. Decreased level and defective function of circulating endothelial progenitor cells in children with moyamoya disease. J Neurosci Res. 2010 Feb 15;88(3):510-8. doi: 10.1002/jnr.22228. PMID 19774676
- [Background] Heeschen C, Aicher A, Lehmann R, Fichtlscherer S, Vasa M, Urbich C, Mildner-Rihm C, Martin H, Zeiher AM, Dimmeler S. Erythropoietin is a potent physiologic stimulus for endothelial progenitor cell mobilization. Blood. 2003 Aug 15;102(4):1340-6. doi: 10.1182/blood-2003-01-0223. Epub 2003 Apr 17. PMID 12702503